CLINICAL TRIAL: NCT06977412
Title: The Application Value of Spectral CT in the Accurate Staging of Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yunnan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KYLX2025-105
Record Dates: First submitted 2025-05-09; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Breast Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The application value of spectral CT in the accurate staging of breast cancer (Experimental): Prospectively collect medical images and clinical data related to breast cancer using Philips Quark CT equipment, and evaluate the diagnostic accuracy and clinical application value in the accurate staging of breast cancer. Patients diagnosed with breast cancer in Yunnan Provincial Cancer Hospital from April 2025 to May 2026 were consecutively included, and after scanning with Philips Quark CT, the TNM stage of breast cancer patients was assessed by two radiologists, and finally statistical analysis was performed.
  Interventions: Diagnostic Test: To explore the value of spectral CT in the diagnosis and treatment of breast cancer

INTERVENTIONS:
Diagnostic Test: To explore the value of spectral CT in the diagnosis and treatment of breast cancer — The CT scan is part of the standard treatment protocol.

SUMMARY:
Spectral CT was used to prospectively collect medical images and clinical data related to breast cancer, evaluate the effect of image quality in the diagnosis of breast cancer, and evaluate the application value in the accurate staging of breast cancer, so as to provide a more accurate clinical basis for diagnosis, promote the development of individualized treatment, and ultimately improve the prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* (a) Chest quark energy spectrum CT examination was performed within 1 week before treatment
* (b) Age ≥ 18
* (c) Suspected breast cancer patients
* (d) Patients who signed informed consent

Exclusion Criteria:

* (a) Severe cardiac, pulmonary and renal insufficiency
* (b) Allergic to iodine contrast media
* (c) Unable to cooperate to complete CT examination
* (d) Quark spectrum CT image is poor and cannot be used
* (e) Male, pregnant and lactating female
* (f) Combined with other tumor history
* (g) Incomplete clinical and pathological data
* (h) Pathologically confirmed non breast cancer

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Pathological TNM staging | 1 day
  Pathological examination information: The pathology results using surgery/biopsy data are the gold standard, and the depth of tumor invasion, lymph node metastasis, and distant metastasis are recorded

CONTACTS AND LOCATIONS:
Overall Officials: Lianhua Ye, Study Director — Ethics Committee of Yunnan Provincial Cancer Hospital